CLINICAL TRIAL: NCT06092671
Title: Effect of Family-centred Perioperative Care for Anaesthesia on Incidence of Emergency Delirium in Children After Surgery: a Protocol for a Randomised Controlled Trial
Brief Title: Effect of FPCA on Incidence of Emergency Delirium in Children After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Jinhua Municipal Central Hospital (Other); Lishui Country People's Hospital (Other); Ningbo No.2 Hospital (Other); The Central Hospital of Lishui City (Other)
Responsible Party: Principal Investigator, TING LI, Principal Investigator, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2023-03-110
Record Dates: First submitted 2023-09-24; First posted 2023-10-23 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Complications; Child; Family; Emergence Delirium; General Anaesthesia; Perioperative Care
Keywords: perioperative care; emergency delirium; paediatric; general anaesthesia; postoperative maladaptive behaviours
MeSH Terms: conditions — Postoperative Complications; Emergence Delirium | interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-Centered group (F group) (Experimental): Both children and parents received family-centred perioperative care for anaesthesia including video education, anaesthesia mask practice, e-manual learning,etc. It is also recommended that a parent accompany the child during both anesthesia induction and recovery.
  Interventions: Other: Family-centred perioperative care for anaesthesia
- Routine group (R group) (No Intervention): The child received clinical standard preoperative education and anesthesia induction. The child was not accompanied by the parents during the anesthesia induction period and the awakening period.

INTERVENTIONS:
Other: Family-centred perioperative care for anaesthesia — The patient in intervention group and parent will receive the Family-centred perioperative care for anaesthesia, including video education, anaesthesia mask practice, electronic pamphlet,etc. It is recommended that parents accompany the children during the induction of anesthesia and the recovery from anesthesia.
  Arms: Family-Centered group (F group)

SUMMARY:
Emergence delirium (ED) stands out as a prevalent postoperative complication among paediatric patients, correlating with extended hospitalization periods, escalated healthcare expenses, and increased incidence of postoperative maladaptive behaviours (POMBs). There is a lack of well-established pharmacological or non-pharmacological interventions demonstrating efficacy in reducing the occurrence of ED. Therefore, our objective is to assess the potential of family-centred perioperative care for anaesthesia (FPCA) in mitigating the incidence of ED in children, compared with routine anaesthesia.

ELIGIBILITY:
Inclusion criteria:

1. Children aged 2-6 years undergoing elective surgery with an estimated surgical duration of no longer than 2 hours;
2. Receiving first general anaesthesia by inhalation, and American Society of Anaesthesiology (ASA) physical status I to II;
3. A parent signed the informed consent form.

Exclusion criteria:

1. Suffering important organ diseases;
2. History of developmental retardation, neuropsychiatric diseases, psychological or cognitive impairment;
3. History of severe hearing or visual impairment;
4. Children are not suitable for inhalation anaesthesia considered by the researchers;
5. The parent involving in this trial spends less than three months a year with the child;
6. The parent is not competent for companionship considered by the researchers;
7. Neither father nor mother is able to participate in the screening interview and the trial.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 444 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of emergency delirium | At the time patient awake from anesthesia after the sugery; 5min after awake; 15min after awake; 25min after awake;
  The incidence of emergency delirium will be evaluated by the Pediatric Anesthesia Emergency Delirium scale (PAED). When the child wakes up in the PACU (the child can stay awake for more than 10 seconds), and 5min, 15min, 25min after waking up, a trained researcher will evaluate the PAED score (the maximum scores ≥10 will be diagnosed as ED).

SECONDARY OUTCOMES:
The severity of emergency delirium | At the time patient awake from anesthesia after the sugery; 5min after awake; 15min after awake; 25min after awake;
  The severity of emergency delirium was assessed according to PAED scores in those patients who suffered emergency delirium. A total score ≥12 is considered moderate emergency delirium, ≥15 is considered severe emergency delirium, and the total score of the scale is 20.
The incidence of postoperative maladaptive behaviours | at postoperative days 1, 2, 3, 7±2, 14±3 days and 3 months ±5 days after surgery
  Postoperative maladaptive behavioural changes at the 1, 2, 3, 7±2, 14±3 days and 3 months±5 days after surgery will be assessed with Post Hospitalization Behaviour Questionnaire (PHBQ). When total score greater than 0 will be considered as postoperative maladaptive behaviours.
Sleep quality | Baseline before surgery; at 7±2, 14±3 days and 3 months ±5 days after surgery
  Sleep quality before surgery and at 7±2, 14±3 days and 3 months ±5 days after surgery, assessed with Children's Sleep Habits Questionnaire (CSHQ).
Quality of life score | Baseline before the surgery and at 14±3 days and 3 months ±5 days after surgery.
  Quality of life score will be assessed with Pediatric Quality of Life Inventory 4.0 (PedsQL4.0).
Compliance of anaesthesia induction | The period anaesthesia induction.
  Compliance of anaesthesia induction in children will be assessed with Induction Compliance Checklist (ICC).
Postoperative pain score | At the time patient awake from anesthesia after the sugery; 5min after awake; 15min after awake; 25min after awake.
  Postoperative pain score in children will be assessed with Face, Legs, Activity, Cry, Consolability scale (FLACC).
Preoperative anxiety of children | Baseline before surgery, in the preoperative holding area and during induction of anaesthesia.
  Preoperative anxiety of children will be assessed with the modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF).
Preoperative anxiety of parents | Baseline before surgery, in the preoperative holding area and during induction of anaesthesia.
  Preoperative anxiety of parents will be assessed with State Trait Anxiety Inventory (STAI).

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, MD. PhD, Principal Investigator — Department of Anaesthesiology and Perioperative Medicine, The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication with no end date
Access Criteria: De-identified participant data underlying the findings will be made available upon reasonable request. Proposals for data access should be directed to the corresponding author (liting1021@aliyun.com).
URL: https://www.wzhealth.com/

REFERENCES:
- [Derived] Chen J, Hu J, Zheng C, Song S, Yang C, Ye F, Li T. Effect of family-centred perioperative care for anaesthesia on the incidence of emergence delirium in children after surgery: a protocol for a randomised controlled trial in China. BMJ Open. 2025 Jul 6;15(7):e089863. doi: 10.1136/bmjopen-2024-089863. PMID 40623754